CLINICAL TRIAL: NCT04184895
Title: A Phase 1 Multiple Ascending Intradermal Dose Study to Assess the Safety, Tolerability and Immunological Response of ASP2390 in Adult Subjects Allergic to House Dust Mites
Brief Title: A Study to Assess the Safety, Tolerability and Immunological Response of ASP2390 in Adult Subjects Allergic to House Dust Mites
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2390-CL-0001; 2018-004678-83 (EudraCT Number); 2022-500660-35-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Allergic to House Dust Mites
Keywords: Tolerability; HDM; ASP2390; Safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASP2390 Low Dose (Cohort 1) (Experimental): Participants will receive a low dose of ASP2390 once weekly for a total of 12 doses. After all participants in cohort 1 complete 4 doses of treatment, the overall safety and tolerability of the dose will be evaluated by the Dose Escalation Committee (DEC).
  Interventions: Biological: ASP2390
- Placebo Low Dose (Cohort 1) (Placebo Comparator): Participants will receive a low dose of matching Placebo once weekly for a total of 12 doses.
  Interventions: Biological: Placebo
- ASP2390 High Dose (Cohort 2) (Experimental): Participants will receive a high dose of ASP2390 once weekly for a total of 12 doses. The dose for cohort 2 may be adapted after the DEC evaluates emergent safety and tolerability data.
  Interventions: Biological: ASP2390
- Placebo High Dose (Cohort 2) (Placebo Comparator): Participants will receive a high dose of matching Placebo once weekly for a total of 12 doses.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ASP2390 — Intradermal
  Arms: ASP2390 High Dose (Cohort 2); ASP2390 Low Dose (Cohort 1)
Biological: Placebo — Intradermal; normal saline solution
  Arms: Placebo High Dose (Cohort 2); Placebo Low Dose (Cohort 1)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple ascending intradermal doses of ASP2390 in adult male and female participants allergic to house dust mites (HDM).

This study will also evaluate the effect of multiple ascending intradermal doses of ASP2390 on HDM-specific immunoglobulin G subclass 4 (IgG4) levels in adult male and female participants allergic to HDM.

DETAILED DESCRIPTION:
Screening will occur up to 6 weeks prior to enrollment. Eligible participants will return to the clinical unit on day -1 (if required by the clinical unit to facilitate the severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] real-time reverse transcription polymerase chain reaction [PCR] procedure) or on day 1.

After the first dose on day 1, all participants will remain in the clinical unit for observation for approximately 24 hours postdose. After the 24 hours, participants will be discharged from the clinical unit provided no reactions have occurred that require additional observation.

For all subsequent doses, participants will remain under direct observation for a minimum of 1 hour postdose. Participants will be discharged from the clinical unit provided no reactions have occurred that require additional observation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a history of house dust mite (HDM) induced allergic rhinitis with or without conjunctivitis of 1 year or longer in duration at screening 1.
* Subject has positive skin prick test (SPT) to D. pteronyssinus.
* Subject has a serum specific immunoglobulin E (IgE) level to D. pteronyssinus at screening 1 or within the past 12 months (if performed and documented at the clinical unit).
* Subject shows a positive symptomatic reaction to an HDM based on total nasal symptom score (TNSS) during the challenge test at screening 2.
* Subject has a forced expiratory volume in 1 second (FEV1) of 80% of predicted value or greater at screening 1.
* Subject has a body mass index (BMI) range of 18.5 to 35.0 kg/m2, inclusive and weighs at least 50 kg at screening 1.
* A female subject is eligible to participate if the female subject is not pregnant and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP), OR
  * WOCBP who agrees to follow the contraceptive guidance starting at screening 1 and throughout the initial safety follow-up period.
* Female subject must agree not to breastfeed starting at screening 1 and throughout the initial safety follow-up period.
* Female subject must not donate ova starting at screening 1 and throughout the initial safety follow-up period.
* A male subject with female partner(s) of childbearing potential must agree to use contraception until after completion of the initial safety follow-up period.
* A male subject must not donate sperm until after completion of the initial safety follow-up period.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner(s) is(are) breastfeeding until after completion of the initial safety follow-up period.
* Subject agrees not to participate in another interventional study while receiving study drug in present study and until after completion of the initial safety follow-up period.

Exclusion Criteria:

* Subject with concomitant allergies to seasonal aeroallergens which are anticipated to be or become active through the completion of the week 18 daily symptom diary.
* Subject with a concomitant allergy to an animal dander who has exposure on a regular basis to the respective animal dander.
* Subject has received immunosuppressive treatment within 3 months prior to screening 1.
* Subject has received previous immunotherapy treatment with any HDM allergen within 3 years prior to screening 1.
* Subject is receiving ongoing treatment with any specific immunotherapy for other allergies or plans to receive during the course of the primary study period.
* Subject who has used systemic (or inhaled) steroid, mast cell stabilizing drug, T-helper cell type 2 (Th2) cytokine inhibitor, thromboxane A2 synthesis inhibitor, thromboxane A2 receptor antagonist, β-blocker, α-adrenergic blockers, ergot alkaloids, angiotensin-converting enzyme inhibitors and/or angiotensin-receptor blockers within 2 months prior to first study drug administration.
* Subject who has used biologics that are immune modulators within 3 months prior to first study drug administration.
* Subject who has received or is planning to receive vaccination of a live vaccine within 28 days prior to the first administration of the study drug and/or subject who has received or is planning to receive vaccination of an inactive vaccine/toxoid within 7 days prior to the first administration of the study drug during the primary study period.
* Subject with mild to severe asthma receiving therapy.
* Subject has a nasal condition that could confound the efficacy or safety assessments.
* Subject who has history of allergic reactions such as anaphylactic shock, exanthema generalized, angioedema or hypotension caused by HDM and/or any medical products (including vaccine) in the past.
* Subject who has immune disorders and/or diseases requiring immunosuppressive drugs.
* Subject who was diagnosed with immunodeficiency in the past.
* Subject who is unable to discontinue antihistamines.
* Subject has received investigational study drug within 28 days or 5 half-lives, whichever is longer, prior to screening 1.
* Subject has a known or suspected intolerance to lactose and/or milk products.
* Subject has used any prescribed or nonprescribed drugs in the 2 weeks prior to first study drug administration, except for occasional use of paracetamol, topical dermatological products, hormonal contraceptives or hormone replacement therapy (HRT), beta-2-agonist for treatment of asthma or rescue medications for rhinitis and for conjunctivitis, or the coronavirus disease 2019 (COVID-19) vaccine within 7 days prior to the first study drug administration.
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to screening 1.
* Subject has a history of drinking more than 21 units of alcohol per week (> 14 units of alcohol for female subjects) within 3 months prior to screening 1 or the subject tests positive for alcohol or drugs of abuse
* Subject has had significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to screening 1.
* Other exclusion criteria apply.
* Subject has a positive result for SARS-CoV-2 PCR test prior to the chamber challenge at screening 2 (repeat virus testing performed 4 to 7 days apart with the second PCR test to be performed a maximum of 2 days prior to the chamber challenge at screening 2) or prior to randomization on day 1.
* Subject has clinical signs and symptoms consistent with COVID-19 infection, e.g., fever, dry cough, dyspnea, sore throat, fatigue, muscle or body aches and gastrointestinal symptoms or confirmed infection by appropriate SARS-CoV-2 PCR test within the 4 weeks prior to screening 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to week 63
  AEs will be coded using medical dictionary for regulatory activities(MedDRA). An AE is any untoward medical occurrence in a participant administered a study drug which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with use of a medicinal product whether or not considered related to the medicinal product. Confirmed and suspected SARS-CoV-2 infection and COVID-19 will be recorded as an AE. An AE is considered serious if the event: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of ability to conduct normal life functions; results in congenital anomaly or birth defect; requires inpatient hospitalization (except for planned procedures) or leads to prolongation of hospitalization (except if prolongation of planned hospitalization is not caused by an AE); or other medically important events.
Number of participants with laboratory value abnormalities and/or AEs | Up to week 63
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or AEs | Up to week 63
  Number of participants with potentially clinically significant vital sign values.
Number of participants with 12-lead electrocardiogram (ECG) abnormalities and/or AEs | Up to week 63
  Routine 12-lead ECGs will be taken after the participant has been resting in the supine position for at least 5 minutes. Routine 12-lead ECGs will be taken in triplicate.
Number of participants with subcutaneous immunotherapy systemic reaction events | Up to week 11
  Subcutaneous immunotherapy systemic reaction events will be graded using the World Allergy Organization Subcutaneous Immunotherapy Systemic Reaction Grading System.
  Each grade is based on organ system involved and severity. Organ systems are defined as cutaneous, conjunctival, upper respiratory, lower respiratory, gastrointestinal, cardiovascular and other. A reaction from a single organ system such as cutaneous, conjunctival or upper respiratory, but not asthma, gastrointestinal, or cardiovascular is classified as a grade 1. Symptom(s)/sign(s) from more than 1 organ system or asthma, gastrointestinal, or cardiovascular are classified as grades 2 or 3. Respiratory failure or hypotension with or without loss of consciousness define grade 4 and death grade 5. The grade is determined by the physician's clinical judgement.
Number of participants with specific local reactogenicity events | Up to week 12
  Participants will be asked to record local reactogenicity (pain, tenderness, erythema/redness, Induration/Swelling) on a daily basis for 7 consecutive days after the injection, each treatment will be summarized. Grades range from 1 (mild) to 4 (potentially life-threatening).
Number of participants with specific systemic reactogenicity events | Up to week 12
  Participants will be asked to record systemic reactogenicity (nausea/vomiting, diarrhea, headache, fatigue, myalgia) on a daily basis for 7 consecutive days after the injection, each treatment will be summarized. Grades range from 1 (mild) to 4 (potentially life-threatening).

SECONDARY OUTCOMES:
Change from baseline in immunological response to ASP2390 as assessed by HDM allergen-specific IgG4 levels | Baseline and up to week 24
  The house dust mite (HDM) allergen-specific IgG4 immunological response for all participants will be presented for each treatment by visit using descriptive statistics.
Number of participants with Adverse Events | Up to 5 years
  AEs will be coded using medical dictionary for regulatory activities(MedDRA). An AE is any untoward medical occurrence in a participant administered a study drug which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with use of a medicinal product whether or not considered related to the medicinal product. Confirmed and suspected SARS-CoV-2 infection and COVID-19 will be recorded as an AE. An AE is considered serious if the event: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of ability to conduct normal life functions; results in congenital anomaly or birth defect; requires inpatient hospitalization (except for planned procedures) or leads to prolongation of hospitalization (except if prolongation of planned hospitalization is not caused by an AE); or other medically important events.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (2):
- Germany (2):
  - Site DE49001, Berlin
  - Site DE49002, Hanover

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.